CLINICAL TRIAL: NCT00173355
Title: Retrospective Clinical Outcome Study of Pediatric Dermatofibrosarcoma Protuberans: Single Institutional Experience of Twelve Cases From 1977-2002
Brief Title: Clinical Outcome of Pediatric Dermatofibrosarcoma Protuberans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700618
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-08

CONDITIONS: Soft Tissue Neoplasms
Keywords: pediatric Dermatofibrosarcoma Protuberans
MeSH Terms: conditions — Soft Tissue Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Retrospective review of clinical outcome of pediatric Dermatofibrosarcoma Protuberans (PDFSP) after active invitation

DETAILED DESCRIPTION:
Soft tissue sarcoma was rarely seen in pediatric patients, and pediatric Dermatofibrosarcoma Protuberans (PDFSP) was even rare. To our knowledge, the largest report constituted of 19 cases (five of them had no follow-up (FU) status) (1). So we proposed this retrospective study based on the cancer registry of our hospital. Twelve cases who were diagnosed as DFSP before age of 18 were identified. But all of them had been lost of FU for at least two years. So we will try to contact these patients and asked them to be back to our clinic for routine surveillance (history taking and physical exam and optional local image/chest xray) and quality of life (QoL) evaluation after pathological review if this clinical study was approved (2)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as DFSP before age of 18 after pathological review according to the cancer registry of our hospital

Exclusion Criteria:

* age > 18 at diagnosis

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12
Dates: Start 2005-06; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Rong-Sen Yang, M.D., Ph.D., Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan